CLINICAL TRIAL: NCT06396065
Title: A Randomized, Double-blind, Multi-center, Phase III Study of AK112 or Placebo Combined with Pemetrexed and Carboplatin in Patients with EGFR-mutant Locally Advanced or Metastatic Non-squamous NSCLC Who Have Failed to EGFR-TKI Treatment
Brief Title: Phase III Study of AK112 for NSCLC Patients
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Summit Therapeutics (Industry)
Collaborators: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK112-301 (HARMONi)
Record Dates: First submitted 2024-04-25; First posted 2024-05-02 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Non-Squamous Non-small Cell Lung Cancer
Keywords: NSCLC; EGFR Positive; ivonescimab
MeSH Terms: interventions — Pemetrexed; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AK112 in combination with Pemetrexed and Carboplatin (Experimental): Subjects will receive AK112 Plus Pemetrexed and Carboplatin via intravenous infusion (IV) Q3W, up to 4 cycles. Afterward, AK112 Plus Pemetrexed will be used for maintenance treatment (administered on Day 1 of each cycle, Q3W) up to 2 years.
  Interventions: Drug: AK112 Injection
- Placebo in combination with Pemetrexed and Carboplatin (Active Comparator): Subjects will receive Placebo Plus Pemetrexed and Carboplatin via intravenous infusion (IV) Q3W, up to 4 cycles in treatment periods per the randomization schedule. Afterward, Placebo Plus Pemetrexed will be used for maintenance treatment (administered on Day 1 of each cycle, Q3W) up to 2 years.
  Interventions: Drug: Placebo Injection

INTERVENTIONS:
Drug: AK112 Injection — Subjects will receive AK112 Plus Pemetrexed and Carboplatin via intravenous infusion (IV) Q3W, up to 4 cycles. Afterward, AK112 Plus Pemetrexed will be used for maintenance treatment (administered on Day 1 of each cycle, Q3W) up to 2 years.
  Other Names: Pemetrexed; Carboplatin
  Arms: AK112 in combination with Pemetrexed and Carboplatin
Drug: Placebo Injection — Subjects will receive Placebo Plus Pemetrexed and Carboplatin via intravenous infusion (IV) Q3W, up to 4 cycles in treatment periods per the randomization schedule. Afterward, Placebo Plus Pemetrexed will be used for maintenance treatment (administered on Day 1 of each cycle, Q3W) up to 2 years.
  Other Names: Pemetrexed; Carboplatin
  Arms: Placebo in combination with Pemetrexed and Carboplatin

SUMMARY:
A Randomized, Double-blind, Multi-center, Phase III Clinical Study of AK112 or Placebo Combined With Pemetrexed and Carboplatin in Patients With EGFR-mutant Locally Advanced or Metastatic Non-squamous Non-small Cell Lung Cancer Who Have Progressed on or Following Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR-TKI) Treatment (HARMONi)

DETAILED DESCRIPTION:
The trial will be performed as a randomized, Double-Blind, Multicenter trial to compare Ivonescimab (SMT112 /AK112) Plus Pemetrexed and Carboplatin to Placebo Plus Pemetrexed and Carboplatin in Patients with Locally Advanced or Metastatic Non-Squamous Non-Small Cell Lung Cancer (NSCLC) Harboring. Approximately 420 subjects will be randomized to two treatment arms at the ratio of 1:1. Each enrolled subject will receive an intravenous infusion of the Ivonescimab (SMT112 /AK112)/Placebo Plus Pemetrexed and Carboplatin (Q3W,up to 4 cycles) in treatment periods per the randomization schedule. Afterward, Ivonescimab (SMT112 /AK112)/ Placebo Plus Pemetrexed will be used for maintenance treatment (administered on Day 1 of each cycle, Q3W) up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and voluntarily sign a written informed consent form (ICF), which must be signed before the specified study procedures required for the study are performed.
2. Males or females aged ≥ 18 to ≤ 75 years at the time of signing informed consent. (For patients from North America and Europe, there will be no upper age cutoff)
3. ECOG performance status score of 0 or 1.
4. Expected survival ≥3 months.
5. Histologically or cytology-confirmed, locally advanced (Stage IIIB/IIIC) or metastatic (Stage IV) non-squamous NSCLC (according to TNM staging of lung cancer, 8th edition) that cannot be completely resected by surgery and cannot receive radical concurrent/sequential chemoradiation.
6. EGFR activation mutations that are confirmed by tumor histology or cytology or blood test before enrollment (eg, exon 18 point mutations, exon 19 deletions, exon 20 point mutations, and exon 21 point mutations). Patients must provide a previous EGFR mutation test report, otherwise tumor tissue samples, peripheral blood samples, or pleural fluid samples will need to be collected for EGFR status testing prior to enrollment.
7. Prior treatment with EGFR TKI and treatment failure, meeting any of the following requirements: Progression after treatment with first- or second-generation EGFR TKI, and confirmation of absence of T790M mutation after progression (only for patients enrolled in China). Progression after treatment with a third-generation EGFR TKI (eg, osimertinib, ametinib, vometinib). Note, for North America and Europe patients only.
8. According to RECIST v1.1, there is at least 1 measurable noncerebral lesion.
9. Adequate organ function determined by the following requirements
10. Female patients of childbearing age have a negative serum pregnancy test result within 3 days before the first dose
11. If a female patient of childbearing potential has sex with an unsterilized male partner, the patient must use a highly effective method of contraception from the beginning of screening and must agree to continue using these precautions until 120 days after the last dose of the study drug or until 6 months after the last carboplatin and pemetrexed dose (whichever is longer).
12. If an unsterilized male patient has sex with a female partner of childbearing potential, the patient must use an effective method of contraception from the beginning of screening to day 120 after the last dose or until 6 months after the last carboplatin and pemetrexed dose (whichever is longer). The decision to stop contraception after this time point should be discussed with investigator.

Exclusion Criteria:

1. Histologic or cytopathologic evidence of the presence of a small cell carcinoma component, or a predominantly squamous cell carcinoma.
2. Patients who have received immune checkpoint inhibitors (eg, anti-PD-1/L1 antibodies, anti-CTLA-4 antibodies, anti-LAG-3 antibodies, etc.)
3. Received prior systemic chemotherapy, anti-angiogenic therapy, or more than one prior line of antitumor therapy (other than EGFR inhibitors) for advanced stage (IIIB to IV) NSCLC.
4. Concurrent enrollment in another clinical study, unless it is a noninterventional clinical study or the follow-up period of the interventional study is more than 4 weeks from the last dose of the prior clinical study or more than 5 half-lives of the prior study drug, whichever is shorter.
5. Received EGFR inhibitor therapy within 2 weeks (with the exception of osimertinib to be within 7 days) prior to the first dose; received nonspecific immunomodulatory therapy (eg, interleukin, interferon, thymus peptide, tumor necrosis factor) within 2 weeks prior to the first dose, excluding IL-11 for the treatment of thrombocytopenia; have received Chinese herbal medicines or proprietary Chinese medicines with antitumor indications within 1 week before the first dose.
6. Imaging during the screening period shows that the tumor surrounds important blood vessels or has obvious necrosis and/or cavitation of tumor lesions within the lung parenchyma.
7. Imaging during the screening period shows that the tumor invades the surrounding vital organs and blood vessels, such as the heart and pericardium, trachea, esophagus, aorta, superior vena cava, or patient is at risk of esophageal tracheal fistula or esophageal pleural fistula.
8. Symptomatic metastases of the central nervous system.
9. Malignant tumors other than NSCLC within 3 years before the first dose.
10. Active autoimmune disease requiring systemic therapy (eg, with disease-modifying drugs, corticosteroids, immunosuppressant therapy) within 2 years prior to the first dose (excluding ir AEs due to PD-1/L1 inhibitors). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy (prednisone ≤ 10 mg daily or equivalent) for adrenal or pituitary insufficiency) is permitted.
11. There is a history of major diseases before the first dose
12. History of perforation of the gastrointestinal tract and/or fistula, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection, complicated by chronic diarrhea) within 6 months before the first study drug administration.
13. Patients with >30 Gy of chest radiation therapy within 6 months prior to the first dose, nonthoracic radiation therapy >30 Gy within 4 weeks prior to the first dose, and palliative radiation therapy of ≤30 Gy within 2 weeks prior to the first dose and failed to recover from the toxicity and/or complications of these interventions to NCI CTCAE Grade ≤1 (except hair loss and fatigue). Palliative radiotherapy for symptom control is permitted if it has been completed at least 2 weeks before the first dose, and no additional radiotherapy for the same lesion is planned.
14. Inactivated vaccines are allowed. Patients are excluded if they have received a live vaccine or live attenuated vaccine within 4 weeks prior to the first dose, or if they are scheduled to receive a live vaccine or live attenuated vaccine during the study period.
15. Severe infection within 4 weeks prior to the first dose, including but not limited to comorbidities requiring hospitalization, sepsis, or severe pneumonia; active infection that has received systemic anti-infective therapy within 2 weeks prior to the first dose (excluding antiviral therapy for hepatitis B or C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  Progression-free survival (PFS) assessed by IRC per RECIST v1.1 in the ITT population.
Overall Survival (OS) in the ITT population | Up to 2 years
  Overall Survival (OS) in the ITT population

SECONDARY OUTCOMES:
ORR | Up to 2 years
  Efficacy measures such as overall response rate (ORR) and duration of response (DoR), which is the proportion of subjects with CR or PR by IRRC based on RECIST v1.1
AE | From the subject signs the ICF to 30 days (AE) and 90 days (SAE) after the last dose of study treatment or initiation of other anti-tumor therapy, whichever occurs first,up to 2 years
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), and clinically significant abnormal laboratory results.
Observed concentrations of AK112 | through study completion, an average of 2 years
  The endpoints for assessment of PK of AK112 include serum concentrations of AK112 at different timepoints after AK112 administration
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK112 through 90 days after last dose of AK112, up to 2 years
  The immunogenicity of AK112 will be assessed by summarizing the number of subjects who develop detectable antidrug antibodies (ADAs)
DoR | Up to 2 years
  Duration of response (DoR) which is the proportion of subjects with CR or PR by IRRC based on RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (74):
- United States (43):
  - CBCC Global Research, Bakersfield, California
  - UC San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - UCLA Department of Medicine - Hematology/Oncology, Los Angeles, California
  - Palo Alto Medical Foundation Research Institute, Mountain View, California
  - Providence St. Joseph, Orange, California
  - UC Irvine, Orange, California
  - Sutter Cancer center, Sacramento, California
  - UC DAVIS Comprehensive Cancer Center, Sacramento, California
  - Sharp Memorial Hospital, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - Providence Medical Foundation, Santa Rosa, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Rocky Mountain Cancer Center, Lone Tree, Colorado
  - The Oncology Institute of Hope & Innovation, Fort Lauderdale, Florida
  - University of Miami, Miami, Florida
  - Florida Cancer Associates - Ocala Oncology, Ocala, Florida
  - BRCR Global, Plantation, Florida
  - Florida Cancer Specialists - North, St. Petersburg, Florida
  - BRCR Global, Tamarac, Florida
  - Florida Cancer Specialists -East, West Palm Beach, Florida
  - Hematology/Oncology Clinic - SCRI, Baton Rouge, Louisiana
  - New England Cancer Specialists, Scarborough, Maine
  - American Oncology Partners, Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - HealthPartners Cancer Research Center, Saint Paul, Minnesota
  - New York Oncology/Hematology, Clifton Park, New York
  - NYU Langone Laura and Isaac Perlmutter Cancer Center, New York, New York
  - Mount Sinai, New York, New York
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Zangmeister Cancer Center, Columbus, Ohio
  - Oncology Hematology Care, Fairfield, Ohio
  - Williamette Valley Cancer Institute and Research, Eugene, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Medical University South Carolina, Charleston, South Carolina
  - Baptist Hospital, Memphis, Tennessee
  - Texas Oncology South Austin, Austin, Texas
  - Texas Oncology Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - MD Anderson University of Texas, Houston, Texas
  - Texas Oncology Webster, Webster, Texas
  - Virginia Cancer specialisits, Fairfax, Virginia
  - Compass Oncology, Vancouver, Washington
- Canada (6):
  - Cross cancer Institute, Edmonton, Alberta
  - BC Cancer, Vancouver, British Columbia
  - Lung Cancer Canada, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Allan Blaire Cancer Centre, Regina, Saskatchewan
  - Universite Hospital Laval, Québec
- France (5):
  - CHI Creteil, Créteil
  - Léon Bérard Cancer Center, Lyon, Lyon
  - Hospital Bichat-Claude Bernard, Paris
  - Institut Curie, Paris
  - Gustave Roussy Cancer, Villejuif
- Italy (5):
  - Istituto Nazionale dei Tumori, Milan
  - Instituto Europeo di Oncologia, Milan
  - University Hospital of Parma, Parma
  - Campus Bio-Medico University, Roma
  - Istituto Nazionale Tumori, Regina Elena, Rome
- Spain (13):
  - Hospital Teresa Herrera, A Coruña
  - Vall d'Hebron Institute of Oncology, Barcelona
  - Badalona-Hospital Germans Trias i Pujol, Barcelona
  - omplejo Hospitalario Universitario Insular-Materno Infantil de Gran Canaria, Las Palmas
  - Lucus Augusti University Hospital, Lugo
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Instituto de Investigacion Sanitaria-Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Puerta de Hierro University Hospital, Majadahonda
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Nuestro Senora de Valme, Seville
- United Kingdom (2):
  - The Royal Marsden, London
  - The Christie NHS Foundation Trust, Manchester